CLINICAL TRIAL: NCT04728256
Title: The Effects of Antenatal Interventions With Artistic Content Given to Pregnant Women on Mental Health and Maternal Attachment Levels
Brief Title: The Effects of Antenatal Interventions With Artistic Content Given to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Sibel Kıyak, Assist. Professor, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NecmettinEU_Kiyak
Record Dates: First submitted 2021-01-02; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Antenatal Care; Mental Health
Keywords: Antenatal care; Depression; Diary; Laughter therapy; Maternal attachment; Music listening
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: The study was a nonrandomized study including a control group for which the post-test procedure was performed alone. The measurements were also repeated at intervals for those in the intervention group. The study intervention group was carried out with a total of 50 pregnant women, 25 of whom were controls.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): A six-session antenatal care program included both music listening and laughter therapy, and was designed for those in the study group as a session every week. The program was carried out by arranging a session of music listening for one week and a laughter therapy session over the following week. Also, the notes uttered by pregnants women were discussed at the week laughter listening sessions were performed. Data from the intervention group was collected four times as pretest (after providing informed contest), first-interval measurement (fourth week of the intervention), second-interval measurement (the first month following the birth) and post-test (the third month following the birth).The data were collected through Beck depression Inventery (BDI), Edinburg postpartum depressıon scale EPDS, Brief semptom ınventory(BSI) and maternal attachment scale(MAS) evaluate overall mental health status comprehensively. All participants responded to the questionnaire prepared for the study.
  Interventions: Behavioral: Laughter therapy+Music listening+Keeping diary
- Control group (No Intervention): Mothers receiving standard antenatal care in the prenatal period, giving birth, and having a three-month-old baby constituted the control group. The Control group was created after the procedures were completed for those in the intervention group. Only the post test was applied to the control group.The data were collected through Beck depression Inventery (BDI), Edinburg postpartum depressıon scale EPDS, Brief semptom ınventory(BSI) and maternal attachment scale(MAS) evaluate overall mental health status comprehensively. All participants responded to the questionnaire prepared for the study.

INTERVENTIONS:
Behavioral: Laughter therapy+Music listening+Keeping diary — Laughter therapy was carried out by the researcher as a total of three sessions every 15 days, and each session lasted 30 minutes.
  Participants listened to the types of music that they like (pop, Turkish folk music). In the meeting room in FHC, Two professional artists performed music recitals with a guitar and saz (qopuz) to pregnant women, and pregnant women actively participated in this process. The performance was carried out as three sessions, once every 15 days, and each session took 40 minutes.
  In addition to music listening and laughter therapy, the pregnant women were asked to keep a diary to write down their emotions about their health status, pregnancy and baby. Then, each participant had an opportunity to explain her emotions or replies to the questions during the group therapy sessions every 15 days so that pregnant women were able to express their feelings.
  Arms: İntervention group

SUMMARY:
Aim:This study aimed to evaluate the effects of music listening, laughter therapy, and diary keeping, given as group sessions to pregnant women in the last trimester on mothers' overall mental health and maternal attachment status in the postpartum period.

Method: The study was a nonrandomized study including a control group for which the post-test procedure was performed alone. The measurements were also repeated at intervals for those in the intervention group. The study was conducted in two separate family health centers.The women with the following constituted the study inclusion criteria: Pregnant women over the age of 18, those with pregnancy between 16-24 weeks of gestation, and those with literacy in Turkish. The data were collected through Beck Depression Inventory, Edinburg Postpartum Depression Scale, Brief Symptom Inventory, and the Maternal Attachment Scale to comprehensively evaluate mental health status. All participants responded to the personal information form prepared for the study.

Keywords:Antenatal care, depression, diary, laughter therapy, maternal attachment, music listening

DETAILED DESCRIPTION:
The intervention group consists of pregnant women in the second trimester who were registered with two family health centers.The Gpower 3.1.9.2. program was used to determine the number of participants in both groups. The sample size was found as 25 for each group by accepting the effect size to be wide (0.82), the alpha value (0.05), and the power (0.80). In the experimental group, sampling adequacy for within comparisons was evaluated with Gpower 3.1.9.2. program. It was determined that the sample was sufficient for partial eta squared values obtained from the study. (10 participants were adequate for each group).The researcher (SK) obtained the list of registered women with a pregnancy between 16-24 gestational weeks. Based on the inclusion and exclusion criteria, the participants were included in the intervention group via face-to-face interviews. Informed written consent was obtained from each participant, and the interventions were performed in this group. Mothers receiving standard antenatal care in the prenatal period, giving birth, and having a three-month-old baby constituted the control group. The control group was created after the procedures were completed for those in the intervention group.

Interventions such as music listening, laughter therapy, and diary keeping were carried out for each woman in the intervention group.A six-session antenatal care program included both music listening and laughter therapy and was designed for those in the study group as a session every week. The program was carried out by arranging a music session for one week and a laughter therapy session over the following week. Also, the notes uttered by pregnant women were discussed at the week laughter listening sessions were performed. Data from the intervention group were collected four times as pretest (after providing informed contest), first-interval measurement (fourth week of the intervention), second-interval measurement (the first month following the birth), and post-test (the third month following the delivery). Even so, the post-test was administered only for the controls.

The data pooled after the study were analyzed using the computer software of SPSS 22.0, OpenMeta[Analyst], and JAPS 09.0 statistical analysis packages. The findings were tested at p<0.05 of the significance level.Similarity analyses of the study and control groups were performed with chi-square (the Pearson and Yates correction). The post-test scores of BDI, EPDS, BSI, and MAS in the intervention and control groups were compared through the t test in independent groups, and Cohen's d and confidence interval (CI) was utilized in the assessment of effect size. Four measurement results of the intervention group were compared with those of variance analysis through repeated measurements, and the partial eta square and CI were used to evaluate the effect size. Two-way variance analysis for repeated measurements was used in evaluating the group/time interactions of the changes in terms of the overall mental health scores of the group with and without depression symptoms in the intervention group at the four time-point.In Cohen's d calculation, if d is 0.20, 0.50, and 0.80, the calculation demonstrates small, medium, and large effect sizes, respectively (d≤ 0.20 weak, d<0.50 medium and d≥ 0.80 large effect size). However, in evaluating the partial eta square, 0.01, 0.06, and 0.14 were considered small, medium, and large, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over the age of 18,
* Between 16-24 weeks of gestation,
* Can understand and speak Turkish,
* Pregnant women who agreed to participate in the study after giving information about the study and those with literacy in Turkish.

Exclusion Criteria:

* A psychiatric disorder (through self-reporting),
* The existence of chronic disease for laughter therapy (heart diseases, hypertension, hemorrhoids, urinary incontinence, and epilepsy, etc.),
* Pregnancy with infertility treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 50 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
The Beck Depression Inventory | Change from baseline to 24 weeks
  Mental Health:The Beck Depression Inventory (BDI) is a 21-item self-reporting scale consisting of emotional, cognitive, somatic and motivational components to measure the level and severity changes of depressive symptoms. In BDI, it is seen that as the total score obtained from the scale increases, the individual's level of experiencing depressive emotions increases proportionally. In addition, BDI scores can be classified as minimal depression between 0-9 points, mild depression between 10-16, moderate depression between 17-29, and severe depression between 30-63 points.
  The intervention was applied at 16-24 weeks of gestation and at the 3rd month of postpartum.
Edinburg Postpartum Depression Scale | Change from baseline to 24 weeks
  Mental Health: The Edinburg Postpartum Depression Scale (EPDS) was designed with the aim of screening to determine the risks of depression in pregnancy and postpartum periods. However, EPDS cannot be used to diagnose depression. EPDS is a 4-point likert self-reporting scale and consists of 10 items.
  The intervention was applied at 16-24 weeks of gestation and at the 3rd month of postpartum.
Brief Symptom Inventory | Change from baseline to 24 weeks
  Mental Health:Brief Symptom Inventory was developed to determine the individuals' depression, anxiety, sleep, somatization, obsessive-compulsive disorder and interpersonal sensitivity status as the short form of SCL-90-R Scale.The items are scored between 0 and 4, corresponding to "none" and "too much". BSI has three global indexes as discomfort severity, total symptom and discomfort symptom indexes. The increase obtained from the scores in these indexes demonstrates individuals' negative experiences regarding overall mental health status.
  The intervention was applied at 16-24 weeks of gestation and at the 3rd month of postpartum.
The Maternal Attachment Scale | The third month following the birth
  Maternal Attachment:The Maternal Attachment Scale (MAS) measures the attachment for maternal affection.MAS is a 4-point Likert-type scale with 26 items, each ranging from "always" to "never". The score obtained from the scale varies between 26 and 104.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettineu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No